CLINICAL TRIAL: NCT01627093
Title: Prospective Data Collection of Patients Treated With Proton Therapy for Head and Neck Malignancies
Brief Title: Medical Data Collection of Patients With Head and Neck Cancer Treated With Proton Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA11-0803; NCI-2020-00578 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA11-0803 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, medical chart review): Patients complete questionnaires over 30 minutes before treatment begins, at each visit during treatment, and again at all follow-up visits related to treatment. Patients also have their medical records reviewed.
  Interventions: Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Medical Chart Review — Review of medical records
  Other Names: Chart Review
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial collects medical information from patients with head and neck cancer that have received or are scheduled to receive proton therapy. Collecting and analyzing medical information from patients may provide information on the outcomes and treatment related side effects of proton therapy for head and neck cancer and help doctors improve therapy for future patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the outcomes in patients who have received treatment for their head and neck malignancy with proton radiation therapy.

OUTLINE:

Patients complete questionnaires over 30 minutes before treatment begins, at each visit during treatment, and again at all follow-up visits related to treatment. Patients also have their medical records reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients documented to have head and neck cancer treated with proton therapy at MDACC from January 1, 2008 through April 30, 2012 and patients who receive treatment from May 1, 2012 through December 31, 2018

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients documented to have head and neck cancer treated with proton therapy at MD Anderson Cancer Center in Houston, Texas (MDACC) from January 1, 2008 through April 30, 2012, and patients who receive treatment from May 1, 2012 through December 31, 2018
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2012-01-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival analysis of proton therapy for head and neck malignancies | 7 years
  Retrospective chart analysis will be performed on all patients documented to have head and neck cancer, treated with Proton Therapy at MDACC from January 1, 2008 through April 30, 2012. Prospective chart analysis will be performed on head and neck cancer patients currently being treated at MD Anderson Cancer Center beginning May 1, 2012 through December 31, 2018. Overall survival estimated using Kaplan-Meier method. Cox proportional hazards regression used to explore predictors of time-to-event outcomes. Mann-Whitney test used to compare continuous parameters between temporal cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Frank, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org